CLINICAL TRIAL: NCT03265847
Title: Impact of Culturally-Specific Danger Assessment on Safety, Mental Health and Empowerment
Brief Title: The weWomen and ourCircle Intervention for Immigrant, Refugee and Indigenous Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Arizona State University (Other); University of Maryland, Baltimore (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00062191; 1R01HD081179-01 (NIH)
Record Dates: First submitted 2017-08-21; First posted 2017-08-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Violence, Domestic; Violence-Related Symptom
Keywords: intimate partner violence; safety planning; immigrant, refugee; Native American; risk for future violence; risk for intimate partner homicide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally-tailored Safety Planning (Experimental): Women in the intervention group receive the SDA intervention with the culturally-specific DA integrated as appropriate to the target group (i.e., immigrant, refugee or indigenous).
  Interventions: Behavioral: Culturally-tailored Safety Planning
- Usual Care (No Intervention): The control group receive non-DA informed usual safety planning resources modeled on national and state domestic violence online resources, but not provided with immediate and visual feedback to their level of danger or a tailored safety planning.

INTERVENTIONS:
Behavioral: Culturally-tailored Safety Planning — The intervention will provide safety planning/referrals tailored to the DA
  Arms: Culturally-tailored Safety Planning

SUMMARY:
This study evaluates the impact of administering culturally-specific versions of the Danger Assessment (DA) tool followed by the tailored safety planning/referral via use of internet/smartphone-based safety decision aid (SDA) on immigrant, refugee and indigenous women's empowerment, safety and mental health. Half of survivors will receive tailored safety planning/referral based on their level of risk assessed by the DA, while the other half will receive non-DA informed usual safety planning/referral.

DETAILED DESCRIPTION:
The DA is a tool to assess risk for homicide, near homicide, re-assault or severe re-assault by an intimate partner. In the culturally adapted DA-informed safety decision aid intervention, women answer questions on the DA, receive immediate feedback on their level of danger as well as personalized messages about safety based on their scores on the DA. The risk factors and scores on the DA are then combined with the safety priorities of women to develop a tailored safety action with links to community resources. Using a computerized randomization scheme, women are randomly assigned to either the internet and/or smartphone app accessible SDA website or control website.

This trial is being conducted in various geographical regions in the US to address the following aims:

1. Evaluate the impact of administering culturally adapted DA-informed interactive internet-based SDA intervention on abused women's safety compared to women assigned to the control website. It is hypothesized that at 3, 6, and 12 months post-baseline, the intervention group will have increased safety seeking behaviors and reduced exposure to intimate partner violence in comparison to the control group.
2. Evaluate the impact of administering culturally adapted DA-informed interactive internet-based SDA intervention on abused women's mental health compared to women assigned to the control website. It is hypothesized that at 3, 6, and 12 months post-baseline, the intervention group will have improved mental health in comparison to the control group.
3. Evaluate the impact of administering culturally adapted DA-informed interactive internet-based SDA intervention on promoting abused women's empowerment compared to women assigned to the control website. It is hypothesized that at 3, 6, and 12 months post-baseline, the intervention group will have increased empowerment in comparison to the control group.

The study will establish evidence base for a culturally-informed intervention for immigrant, refugee and indigenous women. The intervention will not only prevent future exposure to intimate partner violence, it will also promote abused women's mental health and empowerment.

ELIGIBILITY:
Inclusion Criteria:

* Experiences of intimate partner violence within the past one year
* Foreign born immigrant or refugee woman OR Native American woman
* 18-64 years of age
* Can access and use internet

Exclusion Criteria:

* No experience of intimate partner violence within the past one year
* US born and not Native American
* Younger than 18 or older than 64
* Cannot access or use internet

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 688 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in severity and frequency of physical violence | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The adapted version of the Revised Conflict Tactics Scale (CTS2; Straus 1996) is used to measure severity and frequency of the abusive or violent acts in intimate partner relationships. The CTS2 subscales include physical aggression, injury, psychological aggression and sexual coercion. Response categories range from 0=never to 6= more than 20 times within the past 12 months; 7 = not in referent period but happened before. Higher values on the measure within the past 12 months indicate severe or more frequent experiences of violence. The CTS-2 items are scored using the severity-times-frequency weighted score, as recommended by Straus.

SECONDARY OUTCOMES:
Change in depressive symptoms | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The Patient Health Questionnaire (PHQ-9) is a 9 item measure to assess past two weeks depression symptoms based on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual (DSM-IV). Each of the 9 items score from 0 (not at all) to 3 (nearly every day). A total score is computed to measure severity of depression by summing the items. Higher scores indicate more severe depression symptoms (1-4=minimal depression, 5-9=mild depression, 10-14=moderate depression, 15-19=moderately severe depression, and 20-27= severe depression).
Change in symptoms of post-traumatic stress disorder (PTSD) | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  Harvard Trauma Questionnaire (16 items) is used to measure symptoms of PTSD derived from the DSM-IIR/DSM-IV criteria for PTSD, with scores ranging from 1 to 4. The items represent intrusion/re-experiencing, avoidance/numbing and hypervigilance/arousal symptom clusters. The scale for each question includes four categories of response: "1=Not at all," "2=A little," "3=quite a bit," "4=extremely," rated 1 to 4. A total score is obtained using the mean of responses to the items. Higher scores indicate more severe PTSD symptoms.
Change in overall empowerment | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The Personal Progress Scale-Revised (PPS-R; Johnson et al., 2005) is a 28 item self-report measure of empowerment designed to assess multiple areas associated with empowerment such as positive self-evaluation, self-esteem, ability to regulate emotional distress, gender-role and cultural identity awareness, self-efficacy, self-care, problem-solving, assertiveness skills, and access to resources. Participants' responses are rated on a 7-point scale ranging from 1 (Almost Never) to 7 (Almost Always). The items are summed to create a total score for empowerment. The range of scores is 28-196 with higher scores indicating a greater degree of empowerment.
Change in empowerment related to safety | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The MOVERS is a 13 item scale that measures empowerment within the domain of safety (e.g., extent to which a participant has developed a set of safety-related goals and a belief in her ability to accomplish them, the extent to which she feels that her efforts to achieve safety trigger new difficulties and extent to which she has knowledge about and access to support). Participants respond to each item using a five-point scale from "never true" to "always true". The scores on the measure are summed and averaged to produce a total score. Higher scores indicate a greater degree of empowerment related to safety.

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn C Campbell, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Refugee Women's Clinic, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data for all primary and secondary outcome measures will only be available to the investigators and research team members of the project.